Association between the Irrigation-Agitation Techniques and Periapical Healing of Large Periapical Lesions: A Randomized Controlled Trial

**Clinical Trial Number: NCT06204887** 

Date: 16.05.2024

## Statistical analysis

Analyses were carried out in the IBM SPSS 25 program. As the first step of the statistical analysis, the normality of the data was checked with the Shapiro–Wilk test. When normality was ensured, the Wilcoxon signed rank test was applied to examine the difference between the means of two dependent groups. ANOVA was used to examine the difference between the means of three or more independent groups. In cases where the data were not normally distributed, the Kruskal–Wallis test was performed. The post hoc Bonferroni correction was used to determine the group or groups that were significantly different.

Pearson's chi-square test was applied to examine the relationships between study groups and sex. The Kruskal–Wallis test was applied to examine the differences between the average ages of the participants in the study groups. Spearman correlations were used to control for the relationships between age and lesion volume measurements obtained at different times and from different study groups. To compare lesion volume measurements according to study group at different measurement times, ANOVA and the Kruskal–Wallis test were applied. Bonferroni correction were performed to compare the groups. Wilcoxon signed rank tests were used to compare lesion volume measurements according to different measurement times in the study groups.

For comparisons of lesion volume measurements at different measurement times in the study groups, assumptions were checked, and Wilcoxon signed-rank tests were used. Analyses were performed with the IBM SPSS 25 (SPSS Inc., Chicago, IL) program. The Pearson chi-square test was used to examine the relationships between study groups and sex. The Spearman correlation test was used to assess the relationships between lesion volume measurements obtained at different times and study group and age.